CLINICAL TRIAL: NCT04701554
Title: EFFECT OF A 16-SESSION QIGONG PROGRAM ON PHYSICAL AND MENTAL HEALTH IN PATIENTS WITH LYMPHOMA: A RANDOMIZED CONTROLLED TRIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consuelo Lourdes Díaz Rodríguez (Other)
Responsible Party: Sponsor-Investigator, Consuelo Lourdes Díaz Rodríguez, Dr. Consuelo Lourdes Díaz Rodríguez, Universidad de Granada
Organization: Universidad de Granada (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 098988974
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A ramdomized controlled trial.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qigong program (Experimental): The experimental group participated in the Qigong program during 2 months, 16 sessions with a total of 16 hours.
  Interventions: Other: Qigong program
- Active comparator group (Active Comparator): The control group received information on healthy lifestyles, physical exercise and dietary recommendations.
  Interventions: Other: Information on healthy lifestyles, physical exercise and dietary recommendations.

INTERVENTIONS:
Other: Qigong program — The intervention group received sixteen sessions lasting one hour with different techniques of diaphragmatic breathing, concentration techniques and exercises with smooth and coordinated musculoskeletal movements. The Qigong program was performed by a therapist with more than 10 years of experience.
  Arms: Qigong program
Other: Information on healthy lifestyles, physical exercise and dietary recommendations. — The control group received information on healthy lifestyles, physical exercise and dietary recommendations.
  Arms: Active comparator group

SUMMARY:
The aim of the present study was to investigate in lymphoma patients the effects of a 16-session qigong programme (2 times a week) on physical and psychological parameters.

DETAILED DESCRIPTION:
A randomized controlled trial was conducted (control group = 19; intervention = 20). Initially 50 patients enrolled in this study but only 39 finalized the program. 52% male and 48% female with a mean (SD) age of 44.49 (10.60) years. People who have had previous experiencie in mind body practices were excluded. All the patientes received information about the study and informed consent was obtained from all participants. This study was approved by the CEI-GR (C-9) ethics committee and followed the principies of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older; lymphoma histology graded I to IIIA.

Exclusion Criteria:

* Treatment that modifies the vegetative nervous system activity; people that have previous experience in mind body practices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Anxiety and Depression on the Hospital Anxiety and Depression Scale (HADS) after 2 months. | Baseline and after 2 months.
  Validated self-administered instrument for outpatients that advises on the possible presence of anxiety and depression in any non-psychiatric medical consultation. Describe how the patients feel affective and emotionally during the last week.
  It has 14 items, 7 for each subscale with a scale similar to four points (from 0 to 3). Lower scores reflect better outcomes.
Change from Baseline in Happiness on the Lima happiness questionnaire after 2 months. | Baseline and after 2 months.
  Validated self-administered questionnaire consisting of 27 items, integrated into 4 subscales (positive sense of life, satisfaction with life, personal fulfillment and Joy of life), which refer to the level of happiness or satisfaction that the person has with respect to his life.
  The respondent may be: (1) strongly agree, (2) agree, (3) neither agree nor disagree, (4) disagree or (5) strongly disagree, with any question that arises. According to the total score there are 5 levels of happiness: from 27-87 very low happiness; 88-95 low; 96-110 medium; 111-118 high;119-135 very high.
Change from Baseline in Trial Making Test after 2 months. | Baseline and after 2 months.
  A neuropsychological test of visual attention and task switching where the subject is instructed to connect a set of 25 dots as quickly as possible on a sheet of paper. In the first part of the test, the targets are all numbers from 1 to 25 and the test taker needs to connect them in sequential order; in the second part, the dots go from 1 to 13 and include letters from A to L. The patient must connect the dots in order, alternating letters and numbers, as in 1-A-2-B-3-C in the shortest time possible without lifting the pen from the paper.
  The test can provide information about visual search speed, scanning, speed of processing, mental flexibility, as well as executive functioning.
Change from Baseline in Heart rate variability after 2 months. | Baseline and after 2 months.
  We measured short-term HRV using an accepted method in order to assess the cardiovascular balance (Kappussami 2020).
  We asked participants to lie in a supine position for 10 min of rest with normal breathing (following a metronome at 0.2 Hz) and no external stimulation in a quiet room with a temperature of 22-25 ºC.

CONTACTS AND LOCATIONS:
Locations (1):
- Lourdes Díaz Rodríguez, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided